CLINICAL TRIAL: NCT02770209
Title: Autologous Cell-derived Tissue Engineered Cartilage for Repairing Articular Cartilage Lesions: a Protocol for a Prospective, Randomized, Controlled Clinical Trial
Brief Title: Autologous Cell-derived Tissue Engineered Cartilage for Repairing Articular Cartilage Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Quanyi Guo, Director, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLAGH_002
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Cartilage Diseases
MeSH Terms: conditions — Cartilage Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the experimental group (Experimental): Patients in the experimental group will be treated with the biomimetic cartilage matrix combined with autologous chondrocytes. The entire course of treatment includes two surgeries. The first surgery will be performed to observe articular cartilage damage by arthroscopy and assess treatment potential. If the patient's condition meets the surgical requirement, we will extract cartilage from the fossa intercondylar non-weight-bearing area during the first surgery. Chondrocytes will be in vitro-amplified and inoculated into the cartilage scaffold. The fully prepared seeded scaffold will be implanted into the site of injury during the second surgery.
  Interventions: Biological: biomimetic cartilage matrix + autologous chondrocytes
- the control group (Experimental): Patients in the control group will be subjected to arthroscopic debridement and microfracture surgery.
  Interventions: Procedure: arthroscopic debridement; Procedure: microfracture surgery

INTERVENTIONS:
Biological: biomimetic cartilage matrix + autologous chondrocytes
  Arms: the experimental group
Procedure: arthroscopic debridement
  Arms: the control group
Procedure: microfracture surgery
  Arms: the control group

SUMMARY:
This study is aimed at evaluating the feasibility and effectiveness of a completely natural tissue engineered cartilage, composed of a self-made tissue engineered oriented scaffold and autologous chondrocytes, for repairing articular cartilage damage following injury. And it is also aimed at investigating the safety of tissue engineered cartilage transplantation.

DETAILED DESCRIPTION:
Injured articular cartilage has limited capacity for self repair. Without timely, early and effective treatment, damage to the articular cartilage progressively worsens, resulting in joint swelling, pain and dysfunction. The patient ultimately develops osteoarthritis and will be required to undergo artificial joint replacement. Clinical therapy for cartilage damage includes microfracture surgery and autologous osteochondral transplantation. However, the microfracture technique is limited to small-scale damage, and autologous osteochondral transplantation is hindered by limited supply. With advances in material science, cell biology, biomechanics and bioreactor technology, the new generation of biomimetic tissue engineered osteochondral composites display great potential for the repair of cartilage damage.

Currently, in cartilage tissue engineering, seed cells are derived from autologous or allogeneic chondrocytes, mesenchymal stem cells, embryonic stem cells or pluripotent stem cells. Increasing evidence indicates that bone marrow mesenchymal stem cells can be induced to differentiate into chondrocytes, and these cells have been successfully used in the treatment of large-size bone defects, cartilage lesions and spinal cord injury. The quality and quantity of bone mesenchymal stem cells gradually decrease with age, especially in patients with degenerative diseases. Adipose stem cells and umbilical cord mesenchymal stem cells are abundant and have similar characteristics to bone mesenchymal stem cells, and both of these cell types can be induced to differentiate into chondrocytes. Adipose stem cells and umbilical cord mesenchymal stem cells have been used to repair cartilage defects, but the findings are still preliminary, and these cells cannot be harvested or cultured in large quantities. Furthermore, the use of embryonic stem cells is complicated by ethical considerations. As a consequence, autologous chondrocytes are optimal seed cells for cartilage tissue engineering.

The transplantation of autologous chondrocytes in combination with tissue engineered cartilage scaffolds to repair cartilage damage requires researchers to focus on two major issues, namely, (i) the in vitro amplification of chondrocytes and (ii) the preparation of biocompatible chondrocyte scaffolds. The preparation of chondrocyte scaffolds requires advanced technique, and currently, only the Institute of Orthopedics at the Chinese PLA General Hospital has the capacity to produce acellular cartilage; there is no other source of tissue engineered cartilage scaffolds in China.

A proprietary allogeneic acellular cartilage-oriented scaffold was successfully created by the Cartilage Tissue Engineering Research Group, Institute of Orthopedics, Chinese PLA General Hospital (with intellectual property rights). The innovative scaffold simulates the composition and spatial structural characteristics of normal cartilage. The preparation methods are as follows: articular cartilage is pulverized to obtain natural cartilage extracellular matrix, which is identical in biochemical composition to extracellular matrix of natural articular cartilage. Then, a porous sponge-like scaffold is prepared using the freeze-drying technique. In vitro experiments and large-animal articular cartilage injury repair experiments have produced good results. Using this material, our research group prepared biomimetic cartilage tissue engineered scaffolds, which mimic the structural characteristics of natural articular cartilage extracellular matrix. This allogeneic acellular cartilage scaffold has the following characteristics: (1) it is derived from allogeneic cartilage, and the extracellular matrix remains intact after allografting, helping to maintain the numerous components of normal cartilage, particularly type II collagen and proteoglycans, resulting in enhanced repair. Cartilage scaffolds used outside of China are mainly composed of types I and III collagen or hyaluronic acid, and vary greatly from natural cartilage components. The original cartilage structure is difficult to reproduce with these types of scaffolds, and fibrous cartilage may affect treatment outcome. (2) The biomimetic scaffold has a similar three-dimensional structure to that of normal articular cartilage, which is the oriented scaffold structure. The scaffold imitates the orientation of normal cartilage cells, which are arranged perpendicular to the surface, and provides a paratactic columnar structure that contributes to the columnar arrangement of cells. This structure in combination with type II collagen and proteoglycans derived from normal articular cartilage results in a scaffold structure that is extremely close to that of normal joint cartilage. Consequently, the repaired cartilage will have normal structure and function. (3) The oriented scaffold has a good biomechanical property. Its compressive stress is better than the non-oriented scaffold in wet and dry conditions. (4) The oriented scaffold has good biocompatibility. Preliminary experiments have investigated the immune responses of the oriented scaffold of heterogeneous (porcine) and conspecific (rabbit) acellular cartilage. After the oriented scaffold was implanted into the rabbit, its immune responses were observed from the aspects of cellular immunity and humoral immunity. Results suggested that its immunogenicity was low. Thus, it is verified that the oriented scaffold of acellular cartilage has good biocompatibility.

Adverse Events

1. Security Standard operating procedures for adverse events and severe adverse events will be developed to ensure that any adverse reactions during the experiment will be treated quickly to protect the participants.
2. Definitions 2.1 Adverse events Adverse medical events may occur after cartilage transplantation or microfracture surgery, but they do not necessarily have a causal relationship with treatment.

   Common adverse reactions after cartilage transplantation include fever, joint pain, swelling and effusion. Common adverse reactions after microfracture surgery include fever, joint pain, joint swelling and effusion.

   2.2 The severity of adverse events Adverse events will be classified into three levels: general adverse events, vital adverse events and severe adverse events.

   2.3 Relationship with tissue engineered cartilage The correlation between adverse events and tissue-engineered cartilage will be categorized into "definitely related", "probably related", "possibly unrelated", "irrelevant" or "undetermined".

   2.4 Severe adverse events All events occurring during the trial requiring hospitalization or prolonged hospitalization, or resulting in disability, or affecting the ability to work, or with a risk of death or life-threatening events will be recorded.
3. Adverse event recording All adverse events during the experiment will be collected until the end of the study.
4. Recording and reporting All adverse events will be recorded by physicians, including description of adverse events, occurrence time, end time, severity, frequency, and treatment record.

   Once a severe adverse event occurs, physicians will not only give necessary treatment, but also truthfully report to the local Food and Drug Administration Bureau and the National Food and Drug Administration Bureau within 24 hours, as well as promptly report to the Ethics Committee. The data, treatment and follow-up results will be noted in the report.
5. Follow-up observation of non-severe and severe adverse events If a patient suffers a non-severe adverse event, the course and outcome will be closely monitored. The course of severe adverse events will be recorded in follow-up reports or summary reports. Patients will also be monitored, and observations will be recorded for a period of 30 days after a seizure.

Statistical Analysis

1. Study hypotheses All hypotheses will be evaluated with two-tailed tests. A value of P < 0.05 will be considered statistically significant. Baseline data comparability will be assessed. Two-tailed statistical analysis will be performed with α = 5%.
2. Number of cases A total of 100 patients will be involved in this study and divided into two groups, with 50 cases in each group.
3. Experimental analysis Experimental data will be analyzed using statistical software, SPSS 22.0. Measurement data will be expressed as the mean ± SD, median, maximum, minimum and quartiles; count data will be presented as a percentage (%). Count data between groups will be compared using chi-square test or Fisher exact test. Measurement data between groups will be compared using t-test. Nonparametric variables between groups will be compared using rank sum test.
4. Statistical analysis Statistical analysis will be performed by professional statisticians who will not be involved in the study. All data will be input and reviewed, and a statistical analysis report will be prepared.

Administration

1. Preservation of articular cartilage Cartilage tissue will be preserved and transported in a 50 mL centrifuge tube containing 8 mL of tissue preservation solution, placed on a test tube rack on top of an ice pack, at 4 °C under sterile conditions. Cartilage tissue will be transferred to the Institute of Orthopedics at the Chinese PLA General Hospital within 12 hours.
2. Chondrocyte culture and preservation Autologous chondrocytes will be cultured and amplified in strict accordance with the standards and requirements of the National Institutes for Food and Drug Control. All images and data will be recorded. Cartilage seed cells will be frozen in liquid nitrogen.
3. Data quality assurance (1) Researchers will fill in a case report form (CRF) accurately. (2) Inspectors will regularly verify that all data recorded are correct and complete, and that they are consistent with original records, and will be quickly transferred to the data administrator. (3) The data administrator will further examine CRF tables and return the form to the researchers. (4) Two data clerks will input duplicate data into a computer database. (5) The two separate sets of data will be compared by computer software, and modified according to the CRF. (6) Quality control: 5% of all case data will be randomly selected for manual checking. If the data error is greater than 0.15%, all the data in the database will be manually checked.

ELIGIBILITY:
Inclusion Criteria:

* Patients with full-thickness cartilage injury in knee and ankle joints
* Patients with normal joint movement and stable joint (without injury or less than 1/3 excision of the meniscus; normal cruciate ligament, lateral and medial collateral accessory ligament, or normal Q angle and patellofemoral joint trajectory after transplantation, or corrected to normal by surgery), without valgus or varus deformity
* Patients 14-50 years of age.
* Patients with focal cartilage defects diagnosed by arthroscopy, Outerbridge III/IV grade, cartilage defect size 2.5-10 cm2, intact articular surface (lower than grade II injury according to Outerbridge classification), one or two lesions in the same joint.
* Patients and their families are informed of the treatment and provide signed informed consent.

Exclusion Criteria:

* Poor health
* Blood diseases
* Topical steroid therapy within three months
* Bleeding tendency
* Drug addiction (including narcotic, anesthetic or alcohol addiction)
* Inflammatory joint disease (specific or non-specific arthritis)
* Contagious viral infection
* Metabolic diseases (gout or rheumatism)
* Body mass index > 30 kg/m2
* Pregnant or lactating women, or planning to become pregnant within 1 year after initial registration
* Psychological mental illness, cannot cope with rehabilitation

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-08 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change of Magnetic resonance imaging(MRI) | Before treatment and month 3, month 6, month 12, month 18 after surgery
  using joint MRI, cartilage thickness and fusion with surrounding normal cartilage and subchondral bone, as well as the presence or absence of articular effusion and subchondral bone edema will be assessed.

SECONDARY OUTCOMES:
Change of Lysholm score | Before treatment and month 3, month 6, month 12, month 18 after surgery
  The Lysholm score is out of a possible 100 points.
Change of 2000 IKDC subjective knee evaluation score | Before treatment and month 3, month 6, month 12,month 18 after surgery
  A higher score indicates better knee function. IKDC score is used to evaluate knee function and symptoms. 100 points represents no restrictions of daily life and sports.
Change of KOOS survey | Before treatment and month 3, month 6, month 12,month 18 after surgery
Change of the VAS pain scale | Before treatment and month 3, month 6, month 12,month 18 after surgery
  Joint pain will be evaluated with the VAS pain scale; 0 = painless, 10 = severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Quanyi Guo, Ph.D, Principal Investigator — Institute of Orthopedics, Chinese PLA Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ma N, Wang H, Xu X, Wan Y, Liu Y, Wang M, Yu W, Dai Y, Peng J, Guo Q, Yu C, Lu S. Autologous-cell-derived, tissue-engineered cartilage for repairing articular cartilage lesions in the knee: study protocol for a randomized controlled trial. Trials. 2017 Nov 6;18(1):519. doi: 10.1186/s13063-017-2251-6. PMID 29110690